CLINICAL TRIAL: NCT06402136
Title: A Randomised, Double-Blind, Placebo-Controlled, First-in-Human Study of Orally Administered 83-0060 to Evaluate the Safety, Tolerability, and Pharmacokinetics of Single and Multiple Ascending Doses of 83-0060 in Healthy Volunteers
Brief Title: Evaluation Safety, Tolerability, and Pharmacokinetics of Single and Multiple Ascending Doses of 83-0060 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Traws Pharma, Inc. (Industry)
Collaborators: Trawsfynydd Therapeutics AU Pty Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 83-0060-0001; CT-2024-CTN-00084-1 (Other: therapeutic goods administration)
Record Dates: First submitted 2024-05-02; First posted 2024-05-07 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Healthy Volunteers Only

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-Blind, Placebo-Controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Single dose level 1 or placebo (Experimental): Dose level 1. SAD study part.
  Interventions: Drug: 83-0060; Drug: Placebo
- Single dose level 2 or placebo (Experimental): Dose level 2. SAD study part.
  Interventions: Drug: 83-0060; Drug: Placebo
- Single dose level 3 or placebo (Experimental): Dose level 3. SAD study part.
  Interventions: Drug: 83-0060; Drug: Placebo
- Single dose level 4 or placebo (Experimental): Dose level 4. SAD study part.
  Interventions: Drug: 83-0060; Drug: Placebo
- Single dose level 5 or placebo (Experimental): Dose level 5. SAD study part.
  Interventions: Drug: 83-0060; Drug: Placebo
- Multiple dose level 1 or placebo (Experimental): Dose level 1. MAD study part.
  Interventions: Drug: 83-0060; Drug: Placebo
- Multiple dose level 2 or placebo (Experimental): Dose level 2. MAD study part.
  Interventions: Drug: 83-0060; Drug: Placebo
- Multiple dose level 3 or placebo (Experimental): Dose level 3. MAD study part.
  Interventions: Drug: 83-0060; Drug: Placebo

INTERVENTIONS:
Drug: 83-0060 — Oral MPro inhibitor
Drug: Placebo — Placebo

SUMMARY:
This is a clinical study aiming to assess pharmacokinetics, pharmacodynamics and preliminary efficacy of 83-0060 in Healthy Volunteers

DETAILED DESCRIPTION:
This is a Phase 1, double-blind, placebo-controlled, dose escalation study to evaluate the safety, tolerability, PK, PD of orally administered 83-0060 in Healthy Volunteers. The study will be conducted in 2 parts: a single ascending dose (SAD) part at up to 5 dose levels and a multiple ascending dose (MAD) part at up to 3 dose levels. Evaluation of dose levels will be conducted in a sequential fashion with lower dose levels evaluated first in the sequence.

ELIGIBILITY:
Inclusion Criteria:

1. Must have given written informed consent before any study-related activities are carried out and must be able to understand the full nature and purpose of the trial, including possible risks and adverse effects.
2. Adult males and females, 18 to 65 years of age (inclusive) at screening.
3. Body mass index (BMI) ≥ 18.5 and ≤ 32.0 kg/m2, with a body weight (to 1 decimal place) ≥ 50.0 kg at screening.

Exclusion Criteria:

1. History or presence of significant cardiovascular, pulmonary, hepatic, renal, haematological, gastrointestinal, endocrine, immunologic, dermatologic or neurological disease, including any acute illness or major surgery within the past 3 months determined by the PI to be clinically significant.
2. History of surgery or hospitalisation within 30 days prior to screening, or surgery planned during the study.
3. Acute infections within 4 weeks prior to screening or current infection that requires systemically absorbed antibiotic, antifungal, antiparasitic or antiviral medications.
4. Presence or history of any abnormality or illness, including gastrointestinal surgery, which in the opinion of the PI may affect absorption, distribution, metabolism or elimination of the study drug.
5. Any history of malignant disease in the last 5 years (excludes surgically resected skin squamous cell or basal cell carcinoma).
6. Any screening laboratory result outside the normal laboratory reference range (as confirmed upon repeated testing) and deemed clinically significant by the PI.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2024-04-15 (Actual); Primary Completion 2024-08-09 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Incidence of AEs | 8 days in SAD part, 17 days for MAD part
  Incidence of Adverse Events observed during the study
Incidence of drug-related AEs | 8 days in SAD part, 17 days for MAD part
  Incidence of Adverse Events observed during the study deemed related to the study drug by the Investigator
Incidence of SAEs | 8 days in SAD part, 17 days for MAD part
  Incidence of Serious Adverse Events observed during the study
Incidence of lab deviations | 8 days in SAD part, 17 days for MAD part
  Incidence of clinically relevant deviations in the clinical laboratory parameters

SECONDARY OUTCOMES:
Plasma concentration | 8 days in SAD part, 17 days for MAD part
  Plasma concentration, ng/mL

OTHER OUTCOMES:
Pharmacodynamics (PD) of single and multiple oral doses of 83-0060 | 24 hours in SAD part, 11 days for MAD part
  Serum PD endpoint

CONTACTS AND LOCATIONS:
Locations (1):
- Scientia Clinical Research, Sydney, Greater Sydney Area, Australia